CLINICAL TRIAL: NCT06416982
Title: Perineal Massage for Increased Comfort During Pessary Examinations: a Cross-over Randomized Controlled Trial
Brief Title: Perineal Massage for Pessary Examinations
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 24-0544
Record Dates: First submitted 2024-05-13; First posted 2024-05-16 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-05

CONDITIONS: Prolapse, Vaginal; Stress Urinary Incontinence; Pessaries; Pain
Keywords: Pessaries; Vaginal prolapse; Stress urinary incontinence; Pain; Conservative management; Perineal massage
MeSH Terms: conditions — Uterine Prolapse; Urinary Incontinence, Stress; Pain

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Masking Description: Participants will be randomized to intervention vs no intervention at the first visit without stratification, then will undergo the opposite intervention at the second visit. While participants cannot be blinded to the intervention, providers performing the pessary checks and providing provider-perceived pain scores will be blinded to the intervention as someone on the research team other than the provider will perform the intervention prior to the pessary check. If there is unexpected breaking of the blind (e.g. participant tells provider which intervention was performed), the provider will report this to the research team and this will be noted in the study results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Perineal massage before pessary examination (Experimental): Participant will undergo 2 minutes of perineal massage with water-based gel prior to the pessary examination.
  This consists of 2 minutes of perineal massage at the external perineum and sides of the vaginal vestibule, as well as internal massage with the thumb, gliding from 4 to 8 o'clock, then tissue stretching technique with one intracavitary finger and other external finger at the 4 o'clock and 8 o'clock positions three times. The massage will be done by trained doctors who are not performing the pessary check.
  Interventions: Other: Perineal massage
- No perineal massage before pessary examination (No Intervention): Participant will not undergo 2 minutes of perineal massage, but will have water-based gel applied to the vaginal introitus and perineum prior to the pessary check.

INTERVENTIONS:
Other: Perineal massage — 2 minutes of perineal massage as described in arm/group descriptions.
  Arms: Perineal massage before pessary examination

SUMMARY:
Pessaries are effective non-surgical devices for reduction of prolapse. However, use of pessaries are limited in some women due to patient discomfort. While lidocaine can be used to improve pessary checks, its use may be limited due to supply chain shortages, lack of insurance coverage, and optimization of resource utilization. More techniques to improve pessary examination comfort are needed. Perineal massage prior to delivery and at the time of active labor has been noted to reduce perineal trauma and perineal discomfort, theoretically by desensitizing the nerve endings in the skin, broadening the vaginal opening, and increasing elasticity of the perineal tissue. Since most discomfort with pessary checks is during removal and insertion through the vaginal introitus, perineal massage may be a beneficial technique that women could potentially learn to improve comfort with pessary checks.

The objective of this study is to examine the effectiveness of perineal massage prior to pessary check in improving comfort of pessary checks for patients using a cross-over randomized controlled trial.

Patients who follow up for pessary checks with the division of Urogynecology at UNC will be approached about participating in this study. The study will involve two clinical visits. At the first visit, the patient will be randomized to 2 minutes of perineal massage with water based gel of the external perineum and sides of the vaginal vestibule, as well as internal massage with the thumb, gliding from 4 to 8 o'clock, then tissue stretching technique with one intracavitary finger and other external finger at the 4 o'clock and 8 o'clock positions three times; versus application of gel to the internal vagina and external vagina without massage. Providers will be blinded to randomization and proceed with pessary check as per normal clinical protocols.

Patients will rate self-reported pain before, during pessary check, and after the pessary check on a VAS scale; and rate whether they would prefer to repeat this method at future visits via Likert scale. Healthcare professionals will also rate perceived patient pain on VAS scale; ease of pessary removal; and note any perineal or introital laceration or abrasion that may occur during the pessary fitting.

At the following visit, patients will be assigned to the group to which they were not initially randomized. Patients and healthcare professionals will again rate pain as described above. Patients will also rank preference for perineal massage using PGI-I.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing routine pessary management by office providers
* Able to provide informed consent (as reported by patient or family member)
* Able to follow up with the UNC Urogynecology office for two consecutive pessary examination

Exclusion Criteria:

* Non-English speaking
* Found to have a condition such as significant vaginal erosion that precludes replacement of pessary after exam
* Unable to undergo massage due to functional or cognitive impediments or significant discomfort during massage
* Regular usage of pain medications for prior pessary checks such as lidocaine, and unwilling to forgo lidocaine for two study visits
* Pessary visit for pain, pessary expulsion, or significant bleeding, as per provider's judgement

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Patient-perceived pain | 3 months
  Change in pain scores during pessary check (removal and replacement) compared to baseline pain score prior to pessary check using a visual analog scale (VAS) pain scale, as reported by the participant. The VAS pain scale is a validated scale that is performed by having the participant place a mark on a 10 cm line from 0 to 10 to indicate severity of pain. 0 indicates no pain, 10 indicates the most severe pain. Distance from 0 to the mark is measured and recorded in millimeters.

SECONDARY OUTCOMES:
Patient satisfaction with perineal massage | 3 months
  Participants will be asked to rate satisfaction with perineal massage on a 5-point Likert scale. The 5-point Likert scale is a psychometric response method where respondents can easily answer questions and state their level of agreement in five points. The 5-point Likert scale consists of the below points: (1) Strongly Disagree; (2) Disagree; (3) Neither Agree nor Disagree; (4) Agree; (5) Strongly Agree.
Patient preference for future perineal massage | 3 months
  Participants will be asked whether they would choose to undergo perineal massage during future visits. Allowed responses will be Yes/No.
Provider-perceived patient discomfort | 3 months
  The provider performing the pessary examination will be asked to rate patient pain before and during the pessary examination (pessary removal and replacement) on a VAS pain scale. The change in pain score during the pessary examination will be compared. The VAS pain scale is a validated scale that is performed by having the provider place a mark on a 10 cm line from 0 to 10 to indicate severity of pain. 0 indicates no pain, 10 indicates the most severe pain. Distance from 0 to the mark is measured and recorded in millimeters.
Provider-perceived ease of pessary removal | 3 months
  Providers will evaluate ease of pessary removal on a scale of 1 to 10 (with 10 being the most difficult). The ease of pessary removal at the time of the intervention visit will be compared.
Perineal and vaginal abrasion | 3 months
  Providers will be asked to note the presence of any perineal or vaginal abrasions that are thought to be due to pessary removal and/or replacement. The proportion of participants who sustain a perineal or vaginal abrasion will be compared.

OTHER OUTCOMES:
Patient discomfort during perineal massage | At the 3 month follow up visit
  Participants will be asked rate discomfort during the perineal massage on a VAS pain scale.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Chu, MD, MSCI, Principal Investigator — University of North Carollina at Chapel Hill
Locations (1):
- UNC Urogynecology, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No